CLINICAL TRIAL: NCT07291258
Title: Long-term Follow-up of the Offspring Born to Mothers With a Solid Organ Transplant
Brief Title: Long-term Follow-up of the Offspring Born to Mothers With a Solid Organ Transplant, Transplantlines Next Generation
Status: Recruiting | Type: Observational
Sponsor: University Medical Center Groningen (Other)
Collaborators: Groningen Transplantation Fund (GTC) (Unknown); Dutch Transplantation Fund (Unknown); Dutch Kidney Foundation (Other); Astellas Pharma Europe B.V. (Industry); Stichting Eerstelijns Diagnostiek Nederland (SEDN) (Unknown)
Responsible Party: Sponsor
Other Study IDs: METc 2023/610; 10768 (Registry Identifier: Panama ID UMCG); NL85646.042.23 (Registry Identifier: ABR number CCMO)
Record Dates: First submitted 2025-09-03; First posted 2025-12-18 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-11

CONDITIONS: Solid Organ Transplantation; Pregnancy; Long-term Follow-up; Kidney Transplant; Liver Transplant; Pancreas Transplant; Heart Transplantation; Lung Transplantation; Offspring, Adult; Children; Cardiovascular Abnormalities; Kidney Disease; Quality of Life
Keywords: Solid organ transplantation; Pregnancy; Offspring; Long-term follow-up; kidney transplantation; liver transplantation; pancreas transplantation; pancreas islet transplantation; Heart transplantation; lung transplantation
MeSH Terms: conditions — Cardiovascular Abnormalities; Kidney Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood sample, first morning urine sample, feces sample
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Background Pregnancy after all types of solid organ transplantation (SOT) is possible, although these have higher risk of pregnancy complications for mother and child, such as preeclampsia and preterm birth. Thus, the development of the unborn child seems to be affected by the transplant and its consequences such as the immunosuppressive medication use. Worldwide data regarding follow-up after birth is scarce. The very limited existing data existing only in young children are reassuring. However, the investigators hypothesize that there are health risks for the children. Given the side effects of the immunosuppressive medication on patients and limited knowledge from animal studies, the investigators particularly expect cardiovascular effects such as hypertension and kidney damage. These develop over a long time-period and lead late to symptoms.

Aims Aim of this study is to gain more insight into the overall health of offspring born after SOT. Primary aim is to assess the cardiovascular health and the presence of kidney disease, and compare these with reference values from the general population or birth cohorts. Secondary aims are the immunological status including the microbiome of the child given the maternal immunosuppressive medication use, and the overall development of the offspring, including qualitative research regarding the quality of life. Third aim is to assess if there are differences in health between offspring born to mothers with a kidney, liver, pancreas (including pancreas islet), heart and lung transplantation (KTx, LiTx, PTx, HTx, LuTx resp.). The investigators also want to establish a biobank for later follow-up research.

Study design This will be a cross-sectional monocenter cohort study. All offspring ≥16 years of age born after KTx or LiTx and all offspring born at any age after PTx, HTx and LuTx in the Netherlands will be eligible for inclusion. The investigators estimate that there will be about 150(-220) participants. Before the study visit, participants will be asked to complete a questionnaire. Participants will be invited for a one-time study visit consisting of physical tests (including ultrasound of the kidneys and a 24-hour ambulatory blood pressure measurement) and biological sample (urine, blood and feces) collection, including sample collection for biobanking. Information about the growth and development of the offspring and, if present, diseases and medication use will be collected from the medical files of the general practitioner and pharmacy (LSP) and from data from the youth healthcare check-ups. As a control group pseudoanonymized data from the Lifelines cohort will be used.

Deliverables To the best of our knowledge, this will be the first study worldwide that will gather and analyze detailed information about the cardiovascular, kidney and immunological health at a later age (≥16 years) in the offspring born to mothers after KTx, LiTx, PTx, HTx and LuTx. This information will be important for the preconceptional counseling of families with a pregnancy wish after transplantation and thereby contribute to the health of women with a SOT. Next to that, find adverse effects of the pregnancy after transplantation on the offspring are found, the investigators expect there will be modifiable factors and/or early screening/interventions that can reduce these risks and thereby contribute to the health of the offspring.

DETAILED DESCRIPTION:
Rationale:

Studies have reported successful pregnancy outcomes with healthy newborns after all types of solid organ transplantations (SOT). A recent systematic review performed by our center focused on the longer term outcomes (>1 year) of the children born after SOT. We found that data regarding longer term follow-up is scarce, limited to younger children and predominately focused on offspring born after kidney transplantation (KTx) and liver transplantation (LiTx). Only five studies reported outcomes on offspring aged >18 years. The limited existing data in young children are reassuring, development and overall health appears to be similar to the general population. However, it is possible that the development of the fetus is affected by the transplantation and its consequences such as the use of the immunosuppressive medication and the increased incidence of the pregnancy complications, whereby important health risks only become apparent later in life. To gain more insight into the overall health of the offspring born solid organ transplantation and to identify possible pre- and perinatal risks for diseases later in life the investigators want to perform a cross-sectional cohort study. To the best of our knowledge, this will be the first study that will gather and analyze detailed information about the cardiovascular, immunological and kidney health at a later age (≥16 years) in the offspring born to mothers after KTx, LiTx, pancreas (including pancreas islet transplantation), heart and lung transplantation (PTx, HTx, LuTx resp.)

Objective:

The primary aim of this study is to assess the cardiovascular and kidney health of the offspring born after SOT in the mother. Secondary aims are the immunological status including the microbiome of the child and the overall development of the offspring. Third, the investigators want to assess if there are differences in health between offspring born to mothers with a KTx, LiTx, PTx, HTx and LuTx. For the offspring aged <16 years of age the aim is to compare their overall health to the general population.

Study design:

This will be a descriptive cross-sectional monocenter cohort study. All offspring ≥16 years of age born after KTx or LiTx and all offspring born at any age after PTx, HTx and LuTx in the Netherlands will be eligible for inclusion. Eligible participants will be identified via previous studies on pregnancy after KTx, LiTx, HTx and LuTx. Participants will be invited for a one-time study visit consisting of questionnaires, physical tests (including ultrasound of the kidneys) and biological sample (urine, blood and feces) collection. Next to that a 24-hour ambulatory blood pressure measurement will be performed in the participants ≥16 years. The biological sample collection will include sample collection for a biobank. The collection will be in line with the Transplantlines Biobank (METc 2014/077) and an amendment to the Transplantlines Biobank is made and specific informed consent for linking the data of Transplantlines and the current study will be obtained from all participants. For all participants it will be emphasized that the invasive test (blood sample) is optional, participants can still participate in the study if they don't want a blood sample taken. For the participants aged <16 years of age no blood, urine and feces sample will be taken, no ultrasound of the kidney will be performed and a dinamap blood pressure measurement instead of a 24-hour measurement will be performed. Furthermore, data on the pregnancy will be used from three recent national studies, data from the PARTOUT network (national working group on pregnancy after renal transplantation), national data collected on pregnancy after LiTx (manuscript in preparation) and national data on pregnancy after HTx and LuTx (manuscript in preparation). National data to be collected on pregnancy after PTx will be identified and collected through our national network with treating physicians. Information about the growth and development of the offspring and, if present, diseases and medication use will be collected from the medical files of the general practitioner and pharmacy (LSP) and from data from the youth healthcare check-ups. Permission to collect this data will be separately mentioned on the IC. As a control group the investigators will evaluate whether reference values and / or data from existing birth cohorts are available. If not, pseudo anonymized data from the Lifelines cohort will be used.

Study population:

The investigators want to include all offspring aged ≥16 years of age born after KTx or LTx in the mother in the Netherlands. Around 165 children after KTx and around 30 children born after LTx will be eligible for inclusion. Because of the scarcity of pregnancies after PTx, HTx and LuTx worldwide, and as a consequence the lack of information about these pregnancies, the investigators want to include all offspring, at any age, born after PTx, HTx or LuTx heart in the Netherlands. Around 5 children born after HTx and around 12 children born after LuTx will be eligible for inclusion, for children born after PTx this number is still unknown, but will be few. In these young participants the focus will be on the overall health of this group in comparison to a control group. Overall data will be compared to reference values and to a control group of healthy adolescents and (young) adults from existing birth cohorts or the Lifelines cohort.

Main study parameters/endpoints:

The primary endpoints of the study focus on the cardiovascular and kidney health which will be assessed by growth charts and developmental information retrospectively collected from the children's health care center, physical tests (weight and height, body fat and water percentage (BIA), waist-hip-ratio, blood pressure, heart rate and ultrasound of the kidneys) and with biological samples (metabolic parameters: glucose, HbA1c, cholesterol, HDL, LDL, triglycerides, as well as kidney functional parameters: albuminuria, estimated GFR, tubular function).

ELIGIBILITY:
Inclusion Criteria:

* Mother with a KTx, LiTx, PTx (including pancreas islet transplantation), HTx or LuTx before pregnancy (including mothers with multiple transplantation types)
* Age ≥16 years for offspring born to mother with a KTx or LiTx

Exclusion Criteria:

* No informed consent
* Non Dutch or English speaking

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: All offspring born after maternal KTx or LiTx and aged ≥16 years in the Netherlands will be eligible for inclusion. All offspring, at any age born after PTx (including pancreas islet transplantation), HTx or LuTx in the Netherlands will be eligible for inclusion. For all participants it will be emphasized that the invasive test (blood sample) is optional, participants can still participate in the study if they don't want a blood sample taken (or if they don't want to participate in another specific part of the study.) Data will be compared to reference values and/or existing birth cohorts, and if applicable, part of the data will be compared to a control group of healthy adolescents and (young) adults from existing birth cohorts or the Lifelines cohort.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2025-10-15 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2028-06 (Estimated)

PRIMARY OUTCOMES:
Growth charts | Retrospective data on the childhood growth from birth up till 6 years of age and lenght and weight at baseline.
  The primary aim is to assess the cardiovascular and renal health of the offspring born after maternal SOT. One of the outcome measures are growth charts during childhood years.
BMI | Baseline
  The primary aim is to assess the cardiovascular and renal health of the offspring born after maternal SOT. One of the outcome measures is the BMI based on height (m) and weight (kg).
Body fat and water percentage as measured with a bio-impednace meter (BIA). | Baseline
  The primary aim is to assess the cardiovascular and renal health of the offspring born after maternal SOT. One of the outcome measures are the body fat and water percentage as measured with a bio-impednace meter (BIA).
waist-hip ratio | Baseline
  The primary aim is to assess the cardiovascular and renal health of the offspring born after maternal SOT. One of the outcome measures are waist-hip-ratio.
Blood pressure | Baseline
  The primary aim is to assess the cardiovascular and renal health of the offspring born after maternal SOT. One of the outcome measures is blood pressure, measured with a 240hour ambulatory measurement.
Ultrasound of the kidneys | Baseline
  The primary aim is to assess the cardiovascular and renal health of the offspring born after maternal SOT. One of the outcome measures is an ultrasound of the kidneys.
Glucose | Baseline
  The primary aim is to assess the cardiovascular and renal health of the offspring born after maternal SOT. One of the outcome measures is the glucose levels.
HbA1c | Baseline
  The primary aim is to assess the cardiovascular and renal health of the offspring born after maternal SOT. One of the outcome measures is the HbA1c.
Cholesterol | Baseline
  The primary aim is to assess the cardiovascular and renal health of the offspring born after maternal SOT. One of the outcome measures is cholesterol (HDL, LDL, triglycerides)
Albuminuria | Baseline
  The primary aim is to assess the cardiovascular and renal health of the offspring born after maternal SOT. One of the outcome measures is albuminuria.
eGFR | Baseline
  The primary aim is to assess the cardiovascular and renal health of the offspring born after maternal SOT. One of the outcome measures is estimated GFR.
Pulse wave velocity (PWV) | Baseline
  The primary aim is to assess the cardiovascular and renal health of the offspring born after maternal SOT. One of the outcome measures is a 24 hour pulse wave velocity (PWV) measurement.
Troponine | Baseline
  The primary aim is to assess the cardiovascular and renal health of the offspring born after maternal SOT. One of the outcome measures is troponine.
creatine kinase | Baseline
  The primary aim is to assess the cardiovascular and renal health of the offspring born after maternal SOT. One of the outcome measures is creatine kinase.
High sensitive CRP | Baseline
  The primary aim is to assess the cardiovascular and renal health of the offspring born after maternal SOT. One of the outcome measures is high sensitive CRP

SECONDARY OUTCOMES:
Antibiotic use | Retrospective, antibiotic use from birth untill study visit (baseline). Subdivided in antibiotic use during childhood (birth untill 18 years of age) and antibiotic use during adult life (18 years of age untill study visit/baseline)
  Secondary aim is the immunological status, assessed by antibiotic use.
Hospital admissions due to infectious disease | Retrospective, hospital admissions from birth until study visit (baseline). Subdivided in admissions during childhood (birth until 18 years of age) and admissions during adult life (18 years of age until study visit/baseline)
  Secondary aim is the immunological status assessed by hospital admissions due to infectious disease.
IgA | Baseline
  Secondary aim is the immunological status assessed by levels of IgA.
IgM | Baseline
  Secondary aim is the immunological status assessed by levels of IgM.
IgG | Baseline
  Secondary aim is the immunological status assessed by levels of IgG
Leukocyte profiles | Baseline
  Secondary aim is the immunological status assessed by quantitaive analyses of leukocyte profiles
School level | Highest education at time of study visit (baseline) and retrospective data on special education during primary school and secondary school.
  Secondary aim is the overall development of the offspring assessed by school level.
Quality of life ("Positive health questionnaire") | Baseline
  Secondary aim is the overall development of the offspring assessed by Quality of Life questionnaire ("positive health questionnaire")
Chronic diseases | Retrospective, presence of a chronic disease from birth until study visit (baseline). Subdivided in chronic disease during childhood (birth until 18 years of age) and chronic disease during adult life (18 years of age until study visit/baseline)
  Secondary aim is the overall development of the offspring assessed by the presence of chronic diseases
Chronic medication | Retrospective, presence of chronic medication use from birth until study visit (baseline. Subdivided in chronic medication use during childhood (birth until 18 years of age) and chronic medication use during adult life (18 years of age until study visit)
  Secondary aim is the overall health of the offspring assessed by the use of chronic medication

OTHER OUTCOMES:
Differences between the offspring born to mothers with a KTx, LiTx, PTx, HTx and LuTx | Analysis of abnormal findings at study visit subdivided into abnormal findings during childhood (until 18 years of age) and abnormal findings at study visit/baseline (one-time visit).
  An aim of the study is to asses whether differences between the health of the offspring born to mothers with a KTx, LiTx, PTx, HTx and LuTx exist. The investigators will analyse if there are differences in the frequency of chronic diseases and chronic medication use. If the investigators find abnormalities in the kidney function or cardiovascular health (primary aim), they will assess if these abnormalities occur more often in one of the transplantation groups.

CONTACTS AND LOCATIONS:
Overall Officials: Margriet F.C. de Jong, MD, PhD, MBA, Principal Investigator — University Medical Center Groningen
Locations (1):
- University Medical Center Groningen, Groningen, Provincie Groningen, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Transplant Pregnancy Registry International (TPRI), 2022 annual report, Gift of Life Institute, Philadelphia, PA.
- [Result] Eisenga MF, Gomes-Neto AW, van Londen M, Ziengs AL, Douwes RM, Stam SP, Oste MCJ, Knobbe TJ, Hessels NR, Buunk AM, Annema C, Siebelink MJ, Racz E, Spikman JM, Bodewes FAJA, Pol RA, Berger SP, Drost G, Porte RJ, Leuvenink HGD, Damman K, Verschuuren EAM, de Meijer VE, Blokzijl H, Bakker SJL. Rationale and design of TransplantLines: a prospective cohort study and biobank of solid organ transplant recipients. BMJ Open. 2018 Dec 31;8(12):e024502. doi: 10.1136/bmjopen-2018-024502. PMID 30598488
- [Result] Slabiak-Blaz N, Adamczak M, Gut N, Grajoszek A, Nyengaard JR, Ritz E, Wiecek A. Administration of Cyclosporine A in Pregnant Rats - the Effect on Blood Pressure and on the Glomerular Number in Their Offspring. Kidney Blood Press Res. 2015;40(4):413-23. doi: 10.1159/000368515. Epub 2015 Jul 27. PMID 26227088
- [Result] Tendron-Franzin A, Gouyon JB, Guignard JP, Decramer S, Justrabo E, Gilbert T, Semama DS. Long-term effects of in utero exposure to cyclosporin A on renal function in the rabbit. J Am Soc Nephrol. 2004 Oct;15(10):2687-93. doi: 10.1097/01.ASN.0000139069.59466.D8. PMID 15466273
- [Result] Lewandowski AJ, Leeson P. Preeclampsia, prematurity and cardiovascular health in adult life. Early Hum Dev. 2014 Nov;90(11):725-9. doi: 10.1016/j.earlhumdev.2014.08.012. Epub 2014 Sep 7. PMID 25209092
- [Result] Lindstrom L, Skjaerven R, Bergman E, Lundgren M, Klungsoyr K, Cnattingius S, Wikstrom AK. Chronic Hypertension in Women after Perinatal Exposure to Preeclampsia, Being Born Small for Gestational Age or Preterm. Paediatr Perinat Epidemiol. 2017 Mar;31(2):89-98. doi: 10.1111/ppe.12346. Epub 2017 Feb 20. PMID 28218407
- [Result] Shah S, Venkatesan RL, Gupta A, Sanghavi MK, Welge J, Johansen R, Kean EB, Kaur T, Gupta A, Grant TJ, Verma P. Pregnancy outcomes in women with kidney transplant: Metaanalysis and systematic review. BMC Nephrol. 2019 Jan 23;20(1):24. doi: 10.1186/s12882-019-1213-5. PMID 30674290
- [Result] Valentin N, Guerrido I, Rozenshteyn F, Pinotti R, Wu YC, Collins K, Shah M, Hershman M, Weisberg I. Pregnancy Outcomes After Liver Transplantation: A Systematic Review and Meta-Analysis. Am J Gastroenterol. 2021 Mar 1;116(3):491-504. doi: 10.14309/ajg.0000000000001105. PMID 33657039
- [Result] Meinderts JR, Prins JR, Berger SP, De Jong MFC. Follow-Up of Offspring Born to Parents With a Solid Organ Transplantation: A Systematic Review. Transpl Int. 2022 Aug 5;35:10565. doi: 10.3389/ti.2022.10565. eCollection 2022. PMID 35992748